CLINICAL TRIAL: NCT06027866
Title: A Mixed Method Prospective Observational Cohort Study to Test Speech Recognition Application for the Voice Impaired (SRAVI) as a Communication Aid for Acute and Critical Care Patients With Tracheostomies.
Brief Title: A Speech Recognition Application as a Communication Aid for Acute and Critical Care Patients With Tracheostomies
Acronym: SRAVI
Status: Completed | Type: Observational
Sponsor: Queen's University, Belfast (Other)
Collaborators: Western Health and Social Care Trust (Other)
Responsible Party: Sponsor
Other Study IDs: B22/04
Record Dates: First submitted 2023-08-22; First posted 2023-09-07 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Tracheostomy; Communication; Acute/Critical Illness
MeSH Terms: conditions — Communication; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tracheostomy patients: All consenting participants will receive access to SRAVI (Speech Recognition Application for the Voice Impaired), a communication aid for speech-impaired patients. SRAVI is a software-based mobile application ('app') and can be downloaded onto any device with a standard forward facing camera (e.g., smartphone, tablet). SRAVI has been registered with the Medical and Healthcare products Regulatory Agency (MHRA) and CE marked for intended use. SRAVI is based on Visual Speech Recognition (VSR) technology. Specifically, the LipRead technology can determine speech by analysing the movements of a user's lips as they speak into a camera.
  Interventions: Device: SRAVI (Speech Recognition Application for the Voice Impaired)

INTERVENTIONS:
Device: SRAVI (Speech Recognition Application for the Voice Impaired) — Speech Recognition Application for the Voice Impaired (SRAVI) is a novel communication aid developed by Liopa (a company formed by Queen's University Belfast (QUB) and the Centre for Security Information Technologies (CSIT), QUB). SRAVI is an application-based lip-reading system, and the application ('app') can be downloaded onto any device with a standard forward facing camera (e.g., smartphone, tablet). When the device is held in front of a patient, it will track lip movement and identify phrases being mouthed.

SUMMARY:
Patients in acute and critical care often undergo a tracheostomy. A tracheostomy is an incision at the front of the neck to insert a breathing tube directly into the airway. The tube sits in place in the airway using an inflated air-filled cuff. This means that no airflow is directed up and out past the vocal cords through the voice box, and speech is not possible. Being unable to speak can cause distress to patients and may place them at an increased risk of harm if they are unable to express their wishes or needs. It can also increase stress for relatives and healthcare staff as they try to understand what patients are trying to say. Usually when patients cannot talk, staff use different items to help, like a pen and paper. A new communication device that runs on a smartphone or tablet has recently been developed. It is for patients with tracheostomies and works by reading lip movements and translating them into words on the device screen.

The aim of this study is to find out if providing adult acute and critical care patients who have a tracheostomy with the use of this lip-reading device could improve how they communicate. This study will include:

1. Using the lip-reading device in acute and critical care to test if it helps patients with tracheostomies to communicate better.
2. Interviews with patients, relatives and focus groups/interviews with staff to find out their views on communication including the use of the new lipreading device.
3. Follow-up with patients approximately 3-months after acute/critical care discharge to complete some further questions about their physical and mental health.

The study will take place in three critical care units and one acute care unit in Northern Ireland and is expected to last 18 months. The study has been funded by the Public Health Agency Research and Development Division.

DETAILED DESCRIPTION:
Study Design: This is a mixed-method, multi-centre prospective observational cohort study to establish the feasibility of SRAVI. Mixed methods include:

* A multi-centre prospective observational cohort study of SRAVI as an addition to usual communication aids.
* Qualitative interviews/focus groups to inform future study design by exploring patients', their significant others and the critical care MDTs' subjective experiences of the study intervention and outcome measures.

Sample size: The investigators aim to recruit a minimum target of 55 patients. For every patient recruited, the investigators anticipate that three qualitative interviews will be undertaken (i.e., with the patient, their significant other, and at least one healthcare professional). Therefore, a feasible target recruitment is 165 participants.

Consent: Written informed consent will be obtained from participants or a personal or professional consultee in accordance with ethical approval.

Data collection: Data will be collected by the investigators and recorded in the study case report form (CRF).

Baseline data

* Inclusion/exclusion criteria and eligibility screen
* Sex
* Age on admission to hospital
* Date of acute/critical care admission
* Admission diagnosis
* Date of tracheostomy insertion during acute/critical care

Daily data collected

* CAM-ICU score (critical care patients only)
* Frequency of SRAVI delivery
* Compliance with SRAVI use
* Adverse events

Feasibility and clinical outcome data collected in acute/critical care

* Screening
* Recruitment rates
* Adverse events
* Delirium (critical care patients only)

Data collected after critical care discharge

• Duration of critical care stay

Data collected during virtual/telephone/in-person follow-up 3 months following acute/critical care discharge:

* Health related quality of life (HRQoL)
* Post-Traumatic Stress Disorder (PTSD)
* Anxiety and depression
* Cognitive status

Data analysis: Descriptive analysis will be used to analyse data from the observational cohort study. Numbers of patients screened, eligible, recruited, consented, and withdrawn from the study will be reported. Baseline demographic and clinical data will be summarised for study participants. Continuous variables will be summarised as mean (standard deviation) and median (interquartile range) and categorical variables will be summarised as number (percent).

Qualitative interviews/focus groups: Interviews/focus groups will be conducted by the investigator. Interview schedules/focus group topic guides will be developed from discussions within the research team, the patient advisory group, and from literature around study participation. The schedules will include a pre-defined list of questions that will be informed by the objectives of the study. The schedule will enable all participants to be asked similar questions and thus permit comparison of themes across each subject during data analysis.

Qualitative data collection: Interviews/focus groups will be audio recorded and professionally transcribed verbatim using an authorised transcription service. All identifying information will be removed prior to analysis. Transcriptions will be reviewed and verified prior to analysis by the research fellow by comparing the audio and written versions to identify errors.

Qualitative analysis: Qualitative data will be subjected to a thematic analysis, using Newell and Burnard's framework. This approach will permit an inductive process of drawing out important data-driven themes and a deductive process relating the major themes that emerge to the pre-defined objectives of the research. A process of constant comparison, reading, and re-reading of the data will enable identification of emerging themes. The process will be facilitated by using a computer-assisted qualitative data software package, NVIVO.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over
* Patients who acquire a tracheostomy in acute/critical care
* Patients can move lips in a way that articulates words
* Able to communicate in English (a current requirement of the technology)

Exclusion Criteria:

-Patient declined consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute/critical care tracheostomy patients
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bronagh Blackwood, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Wellcome-Wolfson Institute for Experimental Medicine Queen's University Belfast, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tracheostomy Patients
Started | 31
Completed | 29
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Tracheostomy Patients
Number analyzed (Participants) | 31
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [48 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Primary admission diagnosis [Count of Participants; unit: Participants]
  Neurological | 11
  Respiratory | 6
  Gastrointestinal | 5
  Cancer | 5
  Infection | 3
  Cardiac | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Using SRAVI at Least Once
Time Frame: From date of study enrolment until SRAVI no longer required by participant (due to return of natural voice) whilst in the study site or participant has been discharged from study site, an average of 8 weeks.
Measure: Number; unit: Participants
Arm/Group | Tracheostomy Patients
Number analyzed (Participants) | 31
Participants | 31

2. Primary Outcome: Number of Words/Phrases Correctly Identified by SRAVI App
Time Frame: From study enrolment until SRAVI no longer required by participant (due to return of natural voice) whilst in study site or participant has been discharged from study site, an average of 8 weeks.
Population: 468 videos were captured by the SRAVI app, of which 135 videos returned the correct word/phrase mouthed by the participant.
Measure: Count of Units; unit: Videos captured
Units Other Than Participants: Videos captured
Arm/Group | Tracheostomy Patients
Number analyzed (Participants) | 31
Number analyzed (Videos captured) | 468
Videos captured | 135

3. Secondary Outcome: Length of Critical Care Stay
Description: Total number of days patient spent in critical care
Time Frame: From critical care admission to critical care discharge, censored at 8-weeks
Population: 26 of 31 participants were recruited from a critical care setting (5 participants were from an acute care setting and thus did not have a critical care LOS).
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tracheostomy Patients
Number analyzed (Participants) | 26
Days | 43.5 [34 to 58]

4. Secondary Outcome: Duration of Hospital Length of Stay
Description: Total number of days patient spent in hospital
Time Frame: From hospital admission to hospital discharge, censored at 3-months
Population: 31 participants were recruited into the cohort study (26 from a critical care setting and 5 from an acute care setting). 2 participants from the critical care setting withdrew from the study and did not use the SRAVI app but did consent to LOS data being included in analysis.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tracheostomy Patients
Number analyzed (Participants) | 31
Days | 66 [43 to 94]

5. Secondary Outcome: Count of Participants With Delirium During Critical Care Stay
Description: Did participants have delirium during their critical care stay?
Time Frame: Assessed twice per shift using the validated delirium screening tool used in each unit from date of study enrolment until SRAVI no longer used or discharge from critical care. Censored at 8-weeks
Population: Of 31 participants recruited into the cohort study, 26 were from a critical care setting were delirium screening was performed (delirium screening was not performed in the acute care setting where 5 patients were recruited). Of these 26 participants, 2 withdrew from the study and thus delirium data was not collected and analysed for these 2 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tracheostomy Patients
Number analyzed (Participants) | 24
Participants | 21

6. Secondary Outcome: Health Related Quality of Life
Description: Measured by the European Quality of Life-5 Dimensions (EQoL-5D) a generic health-related quality of life questionnaire. Respondents describe their current health state in five dimensions: mobility, ability to self-care, ability to undertake usual activities, pain and discomfort, and anxiety and depression. Each dimension has 5 levels: no problems (score of 1), slight problems (score of 2), moderate problems (score of 3), severe problems (score of 4) and extreme problems (score of 5). The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The questionnaire also features a visual analogue scale ranging from 'best imaginable health state' (score of 100) to 'worst imaginable health state' (score of 0).
Time Frame: Three months following acute/critical care discharge
Population: Of 31 participants recruited to the cohort study, 22 were eligible to complete follow-up questionnaires (2 participants withdrew from the cohort study; 3 participants died and 4 participants were censored). Of the 22 eligible participants, 13 completed follow-up questionnaires and 9 were lost to follow-up.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tracheostomy Patients
Number analyzed (Participants) | 13
units on a scale | 65 [40 to 69]

7. Secondary Outcome: Number of Patients Experiencing Symptoms of Anxiety and Depression
Description: The Hospital Anxiety and Depression Scale (HADS) is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscales.
Time Frame: Three months following acute/critical care discharge
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Tracheostomy Patients
Number analyzed (Participants) | 13
Participants | 7

8. Secondary Outcome: Post-traumatic Stress Disorder
Description: The Impact of Events Scale Revised (IES-R) measures severity of Posttraumatic Stress Disorder (PTSD) symptoms. Items are rated on a 5-point scale ranging from 0 ('not at all') to 4 ('extremely'). The IES-R yields a total score (ranging from 0 to 88); higher scores mean worse symptoms.
Time Frame: Three months following acute/critical care discharge
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tracheostomy Patients
Number analyzed (Participants) | 13
units on a scale | 25 [13.5 to 44.5]

9. Secondary Outcome: Cognitive Status
Description: The Montreal Cognitive Assessment-BLIND (MoCA-BLIND) is a test used to detect cognitive decline. The MoCA-BLIND test examines seven domains (executive/visuospatial function, naming, attention, language, abstraction, recall and orientation) of cognitive function with a total of 11 questions with a maximum score of 30. A score of 26 or over is considered to be normal. A score of less than 26 indicates cognitive impairment (worse outcome). Minimum score is 0.
Time Frame: Three months following acute/critical care discharge
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tracheostomy Patients
Number analyzed (Participants) | 13
units on a scale | 18 [17 to 20]

ADVERSE EVENTS:
Time Frame: For duration participant was enrolled on the cohort study, an average of 8 weeks.
Description: Adverse events were classified according to the following categories:
  * Adverse Event
  * Adverse Device Effect (ADE)
  * Serious Adverse Event
  * Serious Adverse Device Effect (SADE)
  * Unanticipated Serious Adverse Device Effect (USADE)
Arm/Group | Tracheostomy Patients
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT06027866/Prot_SAP_000.pdf